CLINICAL TRIAL: NCT06348550
Title: Effect of the Association of Berberine Fitosoma® and Monacolin K MonaKoPure® on Glyco-metabolic Parameters in Dysglycemic and Dyslipidemic Patients. Single-center, Randomized, Double-blind Study.
Brief Title: Effect of the Association of Berberine Fitosoma® and Monacolin K MonaKoPure® on Glyco-metabolic Parameters in Dysglycemic and Dyslipidemic Patients.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Collaborators: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Giuseppe Derosa, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BFMKP 01
Record Dates: First submitted 2024-03-23; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Dyslipidemias; Dysglycemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Active Comparator)
  Interventions: Dietary Supplement: Berberol® K
- Placebo treatment (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Berberol® K — Nutraceutical containing an association of Berberine Fitosoma® and Monacolin K MonaKoPure®
  Arms: Active treatment
Dietary Supplement: Placebo — Placebo
  Arms: Placebo treatment

SUMMARY:
The objective of this study is to evaluate the effectiveness of the association Berberina Fitosoma® and monacolin K MonaKoPure® (Berberol® K supplement) compared to placebo on glucidic and lipid parameters in subjects with fasting blood glucose (FPG) values between 100 and 125 mg/dl and with total cholesterol (TC) values ≥ 200 mg/dl.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the effectiveness of the association Berberina Fitosoma® and monacolin K MonaKoPure® (Berberol® K supplement) compared to placebo on glucidic and lipid parameters in subjects with fasting blood glucose (FPG) values between 100 and 125 mg/dl and with total cholesterol (TC) values ≥ 200 mg/dl.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese subjects [according to body mass index (BMI)]
* Fasting plasma glucose value between 100 and 125 mg/dl, with impaired fasting glucose or impaired glucose tolerance confirmed with oral glucose tolerance test (OGTT)
* Total cholesterol values ≥ 200 mg/dl

Exclusion Criteria:

* Patients with neoplastic and liver diseases, renal failure
* Patients with type 1 or 2 diabetes mellitus
* Pregnant or breastfeeding women
* Hypersensitivity to any of the ingredients
* Therapy with lipid-lowering drugs
* Use of products containing red yeast rice

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Variation of LDL cholesterol | 12 months
  Reduction of LDL-cholesterol after the nutraceutical or placebo intake

SECONDARY OUTCOMES:
Variation of lipid profile | 12 months
  Reduction of total cholesterol, HDL-cholesterol, triglycerides after the nutraceutical or placebo intake
Change in glycemic status | 12 months
  To evaluate the number of subjects changing from impaired fasting glucose or impaired glucose tolerance to type 2 diabetes mellitus

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico S. Matteo Foundation, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No